CLINICAL TRIAL: NCT06644261
Title: Transvaginal Versus Fluoroscopy-guided Trans Gluteal Pudendal Nerve Block for Pudendal Neuralgia and Chronic Pelvic Pain: a Prospective, Noninferiority, Randomized Controlled Trial
Brief Title: Transvaginal Versus Fluoroscopy-guided Trans Gluteal Pudendal Nerve Block for Pudendal Neuralgia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Sean Francis, MD, OBGYN Department Chair, Fellowship Director Urogynecology, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB #24.0319
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Pudendal Neuralgia; Chronic Pelvic Pain Syndrome
MeSH Terms: conditions — Pudendal Neuralgia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Parallel prospective randomized non-inferiority trial with option for cross-over
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patients will be unable to remain masked to treatment intervention. Procedurists will also be unable to remain masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transvaginal pudendal nerve block (Other): Participants in this arm will receive 10 mL bupivacaine injected into bilateral pudendal nerves via transvaginal approach. This is performed by palpating 1 cm superior and medial to the ischial spine. Participants will receive an injection each 2 weeks, for a total of 3 injections over 6 weeks.
  Interventions: Drug: Bupivacaine injection
- Fluoroscopy guided pudendal nerve block (Other): Participants in this arm will receive 5 mL bupivacaine injected into bilateral pudendal nerves via fluoroscopic guided trans gluteal approach. They will receive one injection over the 6-week duration.
  Interventions: Drug: Bupivacaine injection

INTERVENTIONS:
Drug: Bupivacaine injection — Transvaginal: Palpation 1 cm superior and medial to ischial spine to locate pudendal nerve. 22 gauge spinal needle with trumpet will be placed at this location. Upon negative aspiration, 10 mL of 0.25% bupivacaine will be injected bilaterally.
  Fluoroscopic: Anesthesia Pain medicine fluoroscopy guided injection of 5 mL 0.25% bupivacaine bilaterally in the area of the pudendal nerve based on surrounding landmarks

SUMMARY:
Chronic pain affecting the pelvic and urogenital area is a major clinical problem and can have a profound impact on quality of life and health care costs. Pelvic pain arising from entrapment or neuropathy of the pudendal nerve is known as pudendal neuralgia, which results in chronic perineal pain. This pain syndrome is difficult to diagnose and patients with pudendal neuralgia may present to providers with refractory chronic pelvic pain. Pudendal nerve infiltration or pudendal nerve block (PNB) serves as a diagnostic tool and treatment modality for patients with this condition. To date, there are no published randomized controlled trials comparing imaging-guided PNB to transvaginal finger-guided PNB. While one can assume that image-guided nerve blocks will provide better accuracy for injection and potentially better efficacy in pain relief as a result, no published data exists comparing the outcomes and efficacy between modalities.

The purpose of this prospective, non-inferiority, randomized controlled trial is to compare the efficacy of pain relief from bilateral transvaginal finger-guided pudendal nerve block versus bilateral fluoroscopy-guided trans gluteal pudendal nerve block for patients with pudendal neuralgia.

DETAILED DESCRIPTION:
Primary objective:

Determine the efficacy of pain relief comparing the change in Visual Analog Scale (VAS) from baseline to 6 weeks in women randomized to Transvaginal PNB (without imaging) versus Trans gluteal fluoroscopy-guided PNB.

Upon completion of 6-week follow-up, participants will be given the option to crossover to the alternative treatment arm

Secondary Objectives:

Characterize the effect of either pudendal nerve block approach using the following validated questionnaires

* PROMIS-29 (degree of pain intensity and bother across health domains)
* Pain catastrophizing scale (emotional and cognitive impact of pain)
* Short-form McGill (qualitative pain)
* Patient satisfaction with medical care
* Baseline demographics
* Baseline VAS
* Adverse events
* Determine the time to peak pain relief and duration of injection pain relief

ELIGIBILITY:
Inclusion Criteria:

* women >18 years
* English speaking/reading
* Diagnosis of pudendal neuralgia OR chronic pelvic pain with pain in the distribution of the pudendal nerve for 3 months or longer
* Minimum pain/bother score of 4/10
* Desire for pudendal nerve block

Exclusion Criteria:

* Contraindication to pudendal nerve block (examples: skin or vaginal infection, bupivacaine allergy, uncorrected coagulopathy)
* Pregnant or intending to become pregnant during the study
* Pudendal nerve block from any route within the last 3 months
* Major pelvic surgery within the last 3 months (examples: hysterectomy, prolapse repair, midurethral sling)
* Neurologic disease affecting the perineum (examples: spinal cord injury, multiple sclerosis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Absolute change in Visual Analog Scale (VAS) for pain | 6 weeks
  VAS will be obtained at baseline, post-procedure, weekly until 6 weeks, scale is 0-100 mm with higher scores indicated more pain severity

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville Division of Urogynecology and Reconstructive Pelvic Surgery, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No